CLINICAL TRIAL: NCT01779544
Title: Rehabilitation After Lumbar Surgery
Brief Title: Rehabilitation After Lumbar Disc Surgery: Exercise Therapy and Brief Educational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1861
Record Dates: First submitted 2013-01-24; First posted 2013-01-30 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2017-02

CONDITIONS: Prolapse
Keywords: rehabilitation,surgery,brief intervention, exercises
MeSH Terms: conditions — Prolapse; Motor Activity | interventions — Crisis Intervention; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief intervention only (Active Comparator): Brief intervention, an educational model, consists of information
  Interventions: Other: Brief intervention, an educational model
- Exercise group (Active Comparator): Brief educational intervention combined with exercise therapy
  Interventions: Other: Brief intervention, an educational model; Other: Exercise therapy

INTERVENTIONS:
Other: Brief intervention, an educational model — The goal of the the brief intervention is to provide the patient knowledge to reduce uncertainty so that he or she can understand what is important after lumbar disc surgery so that belief in self-efficacy increases.
Other: Exercise therapy — Patients are instructed to do prescribed exercises the first 3 months after surgery, and to log when they do these
  Arms: Exercise group

SUMMARY:
Rehabilitation after lumbar disc surgery (prolapse) focuses on various elements such as endurance, strength, stretching and information. Evidence concludes that it is not harmful to return to activity after lumbar disc surgery, and restrictions to activities after these operations are today more or less nonexistent. Some studies have shown that high intensity programs might be more effective, but they are probably more expensive. In recent years cognitive interventions have received more attention in rehabilitation programs after lumbar disc surgery. The cognitive approach is focused on providing patient knowledge to reduce uncertainty so that he or she can understand what is important after lumbar disc surgery so that belief in self-efficacy increases. A goal of the rehabilitation is to get the patient to resume normal activities. Reviews ask for how much treatment are needed in a rehabilitation program after lumbar disc surgery.

The study will be a randomized clinical trial. The study will compare two different post-operative rehabilitation programs (general information or general information + exercise therapy). Both groups will begin treatment 1 day after surgery. Subjects in exercise therapy group are supposed to continue with exercises 3 months.

In this study the following hypothesis will be studied:

1. Brief intervention, an educational model, alone after lumbar disc surgery do have the same effect on pain in legs and low back as brief intervention, an educational model, combined with exercise therapy.
2. Exercises which are instructed after lumbar disc surgery in a rehabilitation program, are being done by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lumbar disc prolapse with radicular pain
* Age between 18 and 60

Exclusion Criteria:

* Previous lumbar disc surgery (prolapse)
* Spondyloarthritis
* Arthritis
* Systematic disease
* Heart disease
* Does not understand Norwegian language, spoken or in writing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain in the low back and the legs at 6-8 weeks and 1 year postsurgery | Baseline, 6-8 weeks postsurgery and 1 year postsurgery

SECONDARY OUTCOMES:
Disability and beliefs about the condition | Baseline, 6-8 weeks postsurgery and 1 year postsurgery
Change from baseline in Oswestry Disability Index at 6-8 weeks and 1 year postsurgery | Baseline, 6-8 weeks postsurgery and 1 year postsurgery
Change from baseline in Tampa scale of Kinesiophobia (TSK-13) at 6-8 weeks and 1 year postsurgery | Baseline, 6-8 weeks postsurgery and 1 year postsurgery
Change from baseline in Fear-Avoidance Beliefs Questionnaire (physical activity) at 6-8 weeks and 1 year postsurgery | Baseline, 6-8 weeks postsurgery and 1 year postsurgery
Change from baseline in anticipation to return to work at 6-8 weeks postsurgery | Baseline and 6-8 weeks postsurgery postsurgery
Change from baseline in health condition at 6-8 weeks and 1 year postsurgery | Baseline, 6-8 weeks postsurgery and 1 year postsurgery
Change from baseline in health condition rating at 6-8 weeks and 1 year postsurgery | Baseline, 6-8 weeks postsurgery and 1 year postsurgery
Recidive prolapse | 1 year postsurgery

CONTACTS AND LOCATIONS:
Overall Officials: Kari Indrekvam, phd, MD, Study Director — Helse Bergen HF, Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Ortopedisk klinikk, Kysthospitalet i Hagevik, Bergen, Hordaland, Norway